CLINICAL TRIAL: NCT05059340
Title: Normative Study to Explore Point-of-Gaze (POG), Electromyography (EMG) and Elastography Measurement of the Sternocleidomastoid (SCM) Muscle as an Outcome Variable to Track Post-Surgical Outcomes
Brief Title: Study to Explore Post Surgical Outcomes Using Point-of-Gaze, Electromyography and Elastography of the SCM
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/2910
Record Dates: First submitted 2021-08-03; First posted 2021-09-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The side effects following post surgical neck dissection treatment for tumours in the head and neck (HN) region are weakness of the shoulder and neck muscles, numbness and reduced sensation around the neck and shoulder region and a general impact on the participant's overall fitness. While survival has been emphasized as an important outcome, recovery of treatment-related morbidity and return to pre-treatment quality of life (QOL) for participants after cancer treatment is equally important.

Sternocleidomastoid (SCM) muscle functions to turn the head to the left or right. In particular while performing neck dissections, SCM dissection is a common step. The side effects of SCM dissection is a stiff neck or reduced neck movements. To objectively measure the outcome of the SCM muscle function, it is necessary to determine what is the normal range of motion in healthy subjects turning to the left and right to look at objects in a specific location or Point-of gaze (POG) procedure, as well as the Electromyography (EMG) of the SCM during the movement.

In this normative study, 20 healthy subjects will be recruited to perform this POG assessment as well as EMG and Elastography (ETG) testing of the SCM on the left and right side. Outcome measures will include

1. neck range of motion for flexion, side flexion and rotation
2. EMG activation patterns for SCM

2) muscle thickness & stiffness (as determined by grey scale ultrasound (US) and ETG, respectively) of the SCM

The investigators hypothesize that there will not be any significant differences of POG, EMG and ETG measurements between the left and right side of the SCM in healthy subjects.

DETAILED DESCRIPTION:
20 healthy subjects who are staff working in the SGH (Singapore General Hospital) campus, will be recruited for the normative study. Subjects will be recruited through email invitations to participate in the study. Those who meet the inclusion and exclusion criteria will be selected for testing. In order to ensure there are sufficient gender representation in the normative data, the team will select 10 male and 10 female subjects. Consent will be taken from the subjects.

All subjects will have to undergo the following standard tests; Point of gaze (POG) measurement, Electromyography (EMG) and Ultrasound Elastography (ETG) measurement:

1. POG or Point of gaze measurement: This is a non-invasive assessment tool to assess head and neck movement via 3D motion analysis. Neck range of movement will be assessed using a light source together with the 3D motion capture system.

   Participants will be seated in the middle of the room with reflective markers placed on their head and shoulders. The participants will keep their gaze fixed on an object as the starting position in the neutral position. A light source will appear either to the left or right of the neutral position, and the subject will have to detect this light source and indicate to the researcher when they have located the light source. The light source is pre-set at either 60 or 90 degrees diagonally to the left and right of the subjects. The sequence of the light locations is also pre-set for all subjects so that all subjects follow the same sequence to turn either to the left or right, and if it is located 60 or 90 degrees position. Subjects will turn in total, 6 times to the left and 6 times to the right to complete the measurement.

   The 3D motion analyser will capture the neck turning moment in 3 anatomical planes, flexion-extension, lateral flexion, and rotation, relative to the thorax. Angular velocity and acceleration will also be recorded during the movement.
2. Electromyography (EMG) of the SCM during POG testing will be recorded using electrodes on the left and right SCM. The wireless EMG unit Cometa PICO, will be used to record the EMG during POG assessment simultaneously during the movement. This data will be correlated to the range of motion of the neck.
3. Ultrasound Elastography (ETG) measurement:

Stiffness:

Measurement will be performed using Supersonic Ultrasound Machine (Aixplorer; SuperSonic Imagine, Aix-En-Provence, France) that is equipped with a L15-4 high resolution linear transducer with predefined anatomical landmarks. These landmarks are: the height of the hyoid bone (sternocleidomastoid and upper trapezius muscle) and the acromial process for the middle trapezius, the inside border of the rib to the inside edge of the muscle border (for the serratus anterior), medial edge of the medial side of the spine of scapula (for the rhomboid major). The whole SCM will be separated into 3 sections for the measurement of the stiffness of the muscle - Proximal SCM, Mid SCM & Distal SCM. For each section, 3 stiffness measurements will be obtained. This will result in a total of 9 stiffness (elasticity) measurements for each side of the SCM. The average (mean) reading of the 9 measurements will be taken as the final muscle stiffness for analysis. Bilateral SCM will be evaluated.

Thickness (Grey scale):

The full length of the patient's SCM will be physically measured from the mastoid process to the sternal notch. The mid length (measured from the Mastoid Process) will be marked on the skin and scan will be performed at the marked level. The thickness of the SCM muscle will be measured in the transverse and longitudinal planes at the mid-length of the SCM; and the mean thickness score will be used for final analysis. Subjects are scanned in the supine position with head tilted 15 degrees away from the scanned side. This will be performed on the bilateral SCM of the patient.

All POG, EMG and ETG measurements are taken only once with no follow up visits.

The research data will be sent to the Trusted Third Party appointed by the institution for data de-identification prior to data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* BMI between 18 to 34

Exclusion Criteria:

* Individuals who are currently pregnant or breastfeeding.
* Individuals with pain in the neck/shoulder or have a history of shoulder/neck surgery or trauma, or any known shoulder/neck pathology such as rheumatologic disorders, or prior neurological disease affecting the upper extremity such as stroke.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy SGH staff with no previous head or neck injuries.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Neck range of motion for flexion, side flexion and rotation using motion capture system, Qualisys | Immediately after ultrasound scan
  range is measured using 3 D video analysis of motion capture
EMG activation patterns for SCM using Cometa EMG system | Immediately after ultrasound scan
  EMG is recorded using the wireless Cometa EMG system
Muscle thickness & stiffness (as determined by grey scale ultrasound (US) and elastography (ETG) of the SCM) | During the ultrasound scan
  Measured using Ultrasound scanning

CONTACTS AND LOCATIONS:
Overall Officials: Celia Ia Choo Tan, PhD, Principal Investigator — SingHealth Services
Locations (1):
- Singapore General Hospital, Singapore, Singapore